CLINICAL TRIAL: NCT05111626
Title: A Phase 1b/3 Study of Bemarituzumab Plus Chemotherapy and Nivolumab Versus Chemotherapy and Nivolumab Alone in Subjects With Previously Untreated Advanced Gastric and Gastroesophageal Junction Cancer With FGFR2b Overexpression
Brief Title: Bemarituzumab Plus Chemotherapy and Nivolumab Versus Chemotherapy and Nivolumab for FGFR2b Overexpressed Untreated Advanced Gastric and Gastroesophageal Junction Cancer.
Acronym: FORTITUDE-102
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20210098; 2023-505458-16 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-10-29; First posted 2021-11-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Bemarituzumab; AMG 552; 5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6); Nivolumab; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; FGFR2b Overexpression; Capecitabine and Oxaliplatin (CAPOX)
MeSH Terms: conditions — Stomach Neoplasms | interventions — bemarituzumab; Nivolumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b/3 study:
  * Phase 1b (Part 1) is a single-arm open-label study, which will enroll about 20 participants
  * Phase 3 (Part 2) is a randomized double-blind 2-arm study, which will enroll 508 participants
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Safety Lead-in: Bemarituzumab with mFOLFOX6 and Nivolumab (Experimental): Participants will be administered bemarituzumab at different doses with mFOLFOX6 and nivolumab to determine the recommended phase 3 dose (RP3D) based on occurrence of dose-limiting toxicities (DLTs), and on an evaluation of the overall safety, tolerability, and pharmacokinetics (PK).
  Interventions: Drug: Bemarituzumab; Drug: Nivolumab; Drug: Chemotherapy
- Part 2: Bemarituzumab with chemotherapy (mFOLFOX6 or CAPOX) and Nivolumab (Experimental): Participants will be administered bemarituzumab at the RP3D determined from Part 1 in combination with mFOLFOX6 and nivolumab on a 14-day cycle.
  Or participants will be administered bemarituzumab in combination with CAPOX and nivolumab on a 21-day cycle.
  Interventions: Drug: Bemarituzumab; Drug: Nivolumab; Drug: Chemotherapy
- Part 2: Placebo with chemotherapy (mFOLFOX6 or CAPOX) and Nivolumab (Placebo Comparator): Participants will be administered placebo comparator in combination with mFOLFOX6 and nivolumab on a 14-day cycle.
  Or participants will be administered placebo comparator in combination with CAPOX and nivolumab on a 21-day cycle.
  Interventions: Drug: Nivolumab; Drug: Chemotherapy; Other: Placebo

INTERVENTIONS:
Drug: Bemarituzumab — Bemarituzumab will be administered as intravenous (IV) infusion.
  Other Names: AMG 552
  Arms: Part 1 Safety Lead-in: Bemarituzumab with mFOLFOX6 and Nivolumab; Part 2: Bemarituzumab with chemotherapy (mFOLFOX6 or CAPOX) and Nivolumab
Drug: Nivolumab — Nivolumab will be administered as IV infusion.
Drug: Chemotherapy — mFOLFOX6: 5-fluorouracil, leucovorin, and oxaliplatin will be administered as IV infusion.
  OR CAPOX: oxaliplatin will be administered as IV infusion and capecitabine will be administered orally.
Other: Placebo — Placebo will be administered as IV infusion.
  Arms: Part 2: Placebo with chemotherapy (mFOLFOX6 or CAPOX) and Nivolumab

SUMMARY:
The main objective of Part 1 is to evaluate the safety and tolerability of bemarituzumab plus 5-fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) and nivolumab.

The main objective Part 2 is to compare efficacy of bemarituzumab plus chemotherapy (mFOLFOX6 or capecitabine combined with oxaliplatin (CAPOX)) and nivolumab to placebo plus chemotherapy (mFOLFOX6 or CAPOX) and nivolumab as assessed by overall survival.

ELIGIBILITY:
Inclusion Criteria Part 1 and Part 2:

* Adult with unresectable, locally advanced or metastatic (not amenable to curative therapy) histologically documented gastric or gastroesophageal junction adenocarcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Measurable disease or non-measurable, but evaluable disease, according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1)
* Participant has no contraindications to nivolumab and either mFOLFOX6 or CAPOX chemotherapy as per local prescribing information. Participants in Part 1 must have no contraindications to mFOLFOX6. Participants in Part 2 with contraindications to mFOLFOX6 are permitted and may be administered the CAPOX regimen, if no contraindications for this regimen exist. Participants in Part 2 with contraindications to CAPOX are permitted and may be administered the mFOLFOX6 regimen, if no contraindications for this regimen exist
* Adequate organ function as follows:

  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Hemoglobin ≥ 9 g/dL without red blood cell (RBC) transfusion within 7 days prior to the first dose of study treatment
  * Aspartate aminotransaminase (AST) and Alanine aminotransaminase (ALT) <3 x upper limit of normal (ULN) (or < 5 x ULN if liver involvement)
  * Total bilirubin <1.5 x ULN (or < 2 x ULN if liver involvement or Gilbert's disease)
  * Part 1 only: Calculated or measured creatinine clearance (CrCl) of ≥ 50 mL/minute calculated using the formula of Cockcroft and Gault ([140 - Age] × Mass [kg]/[72 × Creatinine mg/dL]) (x 0.85 if female).
* Part 2 only: Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute calculated using the formula of Cockcroft and Gault ([140 - Age] × Mass [kg]/[72 × Creatinine mg/dL]) (x 0.85 if female).
* INR or prothrombin time (PT) < 1.5 × ULN except for participants receiving anticoagulation, who must be on a stable dose of anticoagulant therapy for 6 weeks prior to enrollment

Additional Inclusion Criteria Part 2:

* No prior treatment for metastatic or unresectable disease except for a maximum of

  1 dose of chemotherapy with or without nivolumab; prior adjuvant, neo-adjuvant, and peri-operative therapy is allowed, provided it has been completed more than 6 months prior to the first dose of study treatment
* Fibroblast growth factor receptor 2b (FGFR2b) ≥ 10% 2+/3+ tumor cells (TC) as determined by centrally performed immunohistochemistry (IHC) testing, based on tumor sample either archival (obtained within 6 months/180 days prior to signing pre-screening informed consent) or a fresh biopsy.

Exclusion Criteria:

* Prior treatment with any selective inhibitor of the fibroblast growth factor (FGF)-FGFR pathway
* Known positive human epidermal growth factor receptor 2 (HER2) status
* Untreated or symptomatic central nervous system disease metastases and leptomeningeal disease
* Peripheral sensory neuropathy grade 2 or higher
* Clinically significant cardiac disease
* Other malignancy within the last 2 years (exceptions for definitively treated disease)
* Chronic or systemic ophthalmologic disorders
* Major surgery or other investigational study within 28 days prior to randomization
* Palliative radiotherapy within 14 days prior to randomization
* Abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
* Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experienced DLTs | 28 days
Part 1: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAEs) | Up to 4.5 years
Part 1: Number of Participants Who Experienced One or More Related TEAEs | Up to 4.5 years
Part 1: Number of Participants With Clinically Significant Changes in Vital Signs | Up to 4.5 years
Part 1: Number of Participants With Clinically Significant Changes in Visual Acuity | Up to 4.5 years
Part 1: Number of Participants With Clinically Significant Changes in Physical Examinations | Up to 4.5 years
Part 1: Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | Up to 4.5 years
Part 2: Overall Survival in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Up to 4.5 years

SECONDARY OUTCOMES:
Part 1: Objective Response (OR) | Up to 4.5 years
Part 1: Duration of Response (DoR) | Up to 4.5 years
Part 1: Disease Control Rate (DCR) | Up to 4.5 years
Part 1: Progression Free Survival (PFS) | Up to 4.5 years
Part 1: Overall Survival | Up to 4.5 years
Part 1: Maximum Observed Concentration (Cmax) of Bemarituzumab | Day 1 to up to 4.5 years
Part 1: Area Under the Concentration Time Curve (AUC) of Bemarituzumab | Day 1 to up to 4.5 years
Part 1: Observed Concentration at the End of a Dose Interval (Ctrough) of Bemarituzumab | Day 1 to up to 4.5 years
Part 1: Number of Participants With Anti-Bemarituzumab Antibody Formation | Day 1 to up to 4.5 years
Part 2: PFS in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Up to 4.5 years
Part 2: Overall Survival in All Randomized Participants | Up to 4.5 years
Part 2: PFS in All Randomized Participants | Up to 4.5 years
Part 2: Number of Participants Who Experienced One or More TEAEs | Up to 4.5 years
Part 2: Number of Participants With Clinically Significant Changes in Vital Signs | Up to 4.5 years
Part 2: Number of Participants With Clinically Significant Changes in Visual Acuity | Up to 4.5 years
Part 2: Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | Up to 4.5 years
Part 2: OR | Up to 4.5 years
Part 2: DoR | Up to 4.5 years
Part 2: DCR | Up to 4.5 years
Part 2: Mean Score in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Version 3.0 (QLQ-C30) Individual Scores in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Up to 4.5 years
Part 2: Change From Baseline in EORTC QLQ-C30 Individual Scores in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Baseline to up to 4.5 years
Part 2: Mean Score in Stomach Cancer Related Symptoms Measured by EORTC Quality of Life Questionnaire-Stomach 22 (QLQ-STO22) in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Up to 4.5 years
Part 2: Change From Baseline in Stomach Cancer Related Symptoms Measured by EORTC QLQ-STO22 in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Baseline to up to 4.5 years
Part 2: Mean Score of Visual Analogue Scale (VAS) Scores as Measured by EuroQol 5-dimensional (EQ-5D-5L) in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Up to 4.5 years
Part 2: Change From Baseline of VAS Scores as Measured by EQ-5D-5L in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Baseline to up to 4.5 years
Part 2: Time to Deterioration in Stomach Cancer Related Symptoms Measured by EORTC QLQ-STO22 in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Day 1 to up to 4.5 years
Part 2: Time to Deterioration in Health-Related Quality of Life (HRQoL) Scores in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Day 1 to up to 4.5 years
Part 2: Time to Deterioration in Physical Function Scores in FGFR2b ≥ 10% 2+/3+ Tumor Cell Staining Participants | Day 1 to up to 4.5 years
Part 2: AUC of Bemarituzumab | Day 1 to up to 4.5 years
Part 2: Cmax of Bemarituzumab | Day 1 to up to 4.5 years
Part 2: Ctrough of Bemarituzumab | Day 1 to up to 4.5 years
Part 2: Number of Participants With Anti-Bemarituzumab Antibody Formation | Day 1 to up to 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (348):
- United States (37):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - The Oncology Institute Clinical Research, Cerritos, California
  - Cancer and Blood Specialty Clinic, Downey, California
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - Torrance Memorial Physician Network, Redondo Beach, California
  - Translational Research in Oncology - US Inc, Santa Monica, California
  - Translational Research in Oncology US Inc, Trio Central Pharmacy, Santa Monica, California
  - Olive View-University of California in Los Angeles Medical Center, Sylmar, California
  - Presbyterian Intercommunity Hospital Health Whitter Hospital, Whittier, California
  - Yale New Haven Hospital Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists - Fort Myers, Fort Myers, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Adventist Health System/Sunbelt, Inc d/b/a AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Summit Medical Group, Florham Park, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Gabrail Cancer Center, LLC, Canton, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Saint Lukes University Health Network, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Central-South, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - United States Oncology Regulatory Affairs Corporate Office, The Woodlands, Texas
  - US Oncology Research Investigational Products Center, The Woodlands, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Aurora Health Care Metro Inc, Milwaukee, Wisconsin
- Argentina (12):
  - Cemic, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Centro Medico Austral, Buenos Aires, Distrito Federal
  - Fundacion Ars Medica, San Salvador de Jujuy, Jujuy Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Exelsus Oncologia Clinica, San Miguel de Tucumán, Tucumán Province
  - Fundacion Respirar, Buenos Aires
  - Hospital Italiano, Capital Federal
  - Sanatorio Allende, Córdoba
  - Hospital Privado Universitario de Cordoba, Córdoba
  - Centro Oncologico Riojano Integral, La Rioja
- Australia (5):
  - GenesisCare -North Shore Oncology, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Grampians Health, Ballarat, Victoria
  - Austin Health, Austin Hospital, Heidelberg, Victoria
- Austria (6):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Landeskrankenhaus Feldkirch, Rankweil
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Krankenhaus Wiener Neustadt, Wiener Neustadt
- Belgium (10):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Hopital De Libramont, Libramont
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Algemeen Ziekenhuis Turnhout Campus Sint-Jozef, Turnhout
- Brazil (14):
  - Hospital Haroldo Juacaba - Instituto do Cancer do Ceara, Fortaleza, Ceará
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Sirio Libanes, Brasília, Federal District
  - Personal Oncologia de Precisao e Personalizada, Belo Horizonte, Minas Gerais
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio 12 Hospital de Amor de Barretos, Barretos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Fundacao Antonio Prudente AC Camargo Cancer Center, São Paulo, São Paulo
  - Instituto Coi, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo Octavio Frias de Oliveira Icesp, São Paulo
- Bulgaria (6):
  - Complex Oncology Center - Burgas, Burgas
  - Specialized Hospital for Active Treatment of Oncology - Haskovo EOOD, Haskovo
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Canada (6):
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Research Institute Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier de L Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec
- Chile (7):
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Centro De Estudios Clínicos Suecia SpA, Santiago, Santiago Metropolitan
  - IC La Serena Research, La Serena
  - Centro de Estudios Clinicos SAGA Spa, Santiago
  - Oncovida, Santiago
  - Icegclinic, Santiago
  - Centro de Estudios Clinicos e Investigaciones Medicas CeCim, Santiago
- China (68):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - The first people's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital Affiliated Hospital of Hubei University of Medicine, Shiyan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College Of Hust, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Inner Mongolia Autonomous Region Peoples Hospital, Hohhot, Inner Mongolia
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Changzhi Peoples Hospital, Changzhi, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University Cancer institute and hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Lishui Municipal central Hospital, Lishui, Zhejiang
  - The First Affiliate Hospital of Ningbo University, Ningbo, Zhejiang
- Colombia (5):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Institucion Prestadora de Servicios de Salud Sociedad Médica Rionegro SA Somer SA, Rionegro, Antioquia
  - Sociedad de Oncologia y Hematologia del Cesar, Valledupar, Cesar Department
  - Fundacion Cardiovascular de Colombia, Bucaramanga, Santander Department
  - Fundacion Oftalmologica de Santander - Foscal, Floridablanca, Santander Department
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova nemocnice, Prague
- France (19):
  - Centre Hospitalier Universitaire Amiens Picardie - Hopital Sud, Amiens
  - Centre Hospitalier Regional Universitaire de Besancon, Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Universitaire de Brest - Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Clermont Ferrand, Hopital Estaing, Clermont-Ferrand
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Limoges - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Rene Gauducheau - Institut de Cancerologie de l Ouest, Saint-Herblain
  - Centre Hospitalier Universitaire Nord de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Institut de cancerologie Strasbourg Europe, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (15):
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Haematologisch Onkologische Praxis Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Regional Kliniken Holding Klinikum Ludwigsburg, Ludwigsburg
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitaetsmedizin Mannheim, Mannheim
  - Klinikum der LMU Muenchen, München
  - Klinikum rechts der Isar der TUM, München
  - Universitaetsklinikum der Eberhard Karls Universitaet Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Klinikum der Stadt Wolfsburg, Wolfsburg
- Prince of Wales Hospital / CUHK, Shatin, New Territories, Hong Kong
- Hungary (8):
  - Semmelweis Egyetem, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (14):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Socio Sanitaria Territoriale Papa Giovanni xxiii, Bergamo
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Ente Ospedaliero IRCCS Saverio De Bellis, Castellana Grotte
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Luigi Vanvitelli, Napoli
  - Istituto Nazionale dei Tumori IRCCS Fondazione Giovanni Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Japan (20):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Poland (12):
  - Beskidzkie Centrum Onkologii Szpital Miejski imienia Jana Pawla Drugiego, Bielsko-Biala
  - Narodowy Instytut Onkologii im M Sklodowskiej-Curie Panstwowy Instytut Badawczy Oddzial w Gliwicach, Gliwice
  - Przychodnia Lekarska Komed Roman Karaszewski, Konin
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji, Olsztyn
  - Mazowiecki Szpital Wojewodzki im Sw Jana Pawla II w Siedlcach spzoo, Siedlce
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Uniwersytecki Szpital Kliniczny nr 1 im prof Tadeusza Sokolowskiego Pum w Szczecinie, Szczecin
  - Lux med onkologia sp zoo szpital szamocka, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
  - Mtz Clinical Research powered by Pratia, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Portugal (8):
  - Unidade Local de Saude de Braga, EPE, Braga
  - Unidade Local de Saude do Alto Ave, EPE, Guimarães
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Cuf porto, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
- Romania (7):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Regional de Gastroenterologie si Hepatologie Prof Dr Octavian Fodor, Cluj-Napoca
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (13):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju-si, Jeollabuk-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (16):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Complexo Hospitalario Universitario A Coruna Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (6):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopitaux Universitaires de Geneve, Geneva
  - Onkozentrum Zuerich, Zurich
  - Universitaetsspital Zuerich, Zurich
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Thailand (5):
  - Chulabhorn Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Prince of Songkla Hospital, Songkhla
- United Kingdom (10):
  - Addenbrookes Hospital, Cambridge
  - University Hospital Coventry, Coventry
  - Ninewells Hospital and Medical School, Dundee
  - Royal Free Hospital, London
  - Guys Hospital, London
  - Christie Hospital, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Wainberg ZA, Kang YK, Lee KW, Qin S, Yamaguchi K, Kim IH, Saeed A, Oh SC, Li J, Turk HM, Teixeira A, Hitre E, Udrea AA, Cardellino GG, Sanchez RG, Zahlten-Kumeli A, Taylor K, Enzinger PC. Bemarituzumab as first-line treatment for locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma: final analysis of the randomized phase 2 FIGHT trial. Gastric Cancer. 2024 May;27(3):558-570. doi: 10.1007/s10120-024-01466-w. Epub 2024 Feb 3. PMID 38308771
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com